CLINICAL TRIAL: NCT04370041
Title: Multicenter, Non-randomized Clinical Trial to Reinforce the Current Efficacy and Safety Clinical Data of the Dokimos Plus Aortic Valve
Brief Title: Dokimos Plus Aortic Valve Implant in 80 Patients Diagnosed With a Heart Valve Disease and Requiring Valve Replacement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Swan Medical S. L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DKPLUS2020
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Stenosis; Regurgitation, Aortic
Keywords: Stenosis; Regurgitation, Aortic
MeSH Terms: conditions — Constriction, Pathologic; Aortic Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: This study intends to reinforce the current clinical information regarding safety and efficacy of the Dokimos Plus aortic valve prosthesis in patients over 65 or younger with contraindication for long-term anticoagulation, in which an aortic valve replacement with a bioprosthesis has been indicated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dokimos Plus aortic valve implantation (Experimental): Dokimos Plus aortic valve implantation in all included patients.
  Interventions: Device: Dokimos Plus aortic valve

INTERVENTIONS:
Device: Dokimos Plus aortic valve — Dokimos Plus aortic valve

SUMMARY:
This study intends to reinforce the current clinical information regarding safety and efficacy of the Dokimos Plus aortic valve prosthesis in patients in whom an aortic valve replacement with a bioprosthesis has been indicated.

DETAILED DESCRIPTION:
Multicenter, non-randomized, longitudinal case series clinical trial designed to reinforce the current safety and efficacy clinical data of the Dokimos Plus aortic valve and renew the CE mark.

The study foresees the inclusion of 80 patients recruited prospectively. Patients over 65 who have been diagnosed with a heart valve disease and who require surgical aortic valve replacement, or younger patients who are unsuitable for long-term anticoagulation due to medical contraindications or lifestyle considerations. The study will collect information on the Dokimos Plus aortic valve transvalvular gradient at 6 months and 12 months after the implantation. In addition, patients will be annually followed-up, up to 10 years after implantation.

The objective of the study valve is to improve life expectancy and quality of life of patients with a diseased aortic valve, replacing it with a bioprosthesis that can be safely implanted, with good hemodynamics and long durability.

Clinical studies carried out up to date have shown that the Dokimos Plus aortic valve presents satisfactory clinical and hemodynamic results, similar to those of other bioprothesis available on the market. In addition, the post-marketing surveillance carried out by the manufacturer has not revealed any relevant events regarding the Dokimos Plus aortic valve safety profile.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18
2. Patients with the ability to understand the study requirements, be able to given written informed consent, and be willing and able to comply with the study requirements (including follow-up visits).
3. Patient candidates to an aortic bioprosthesis implantation according to the standard clinical practice guidelines.
4. Patients requiring isolated aortic valve replacement, or in combination with coronary artery bypass surgery and / or in combination with ascending aorta replacement surgery.
5. Women are eligible for the study if: a) are not pregnant or breastfeeding, b) are not of childbearing potential, c) if women of childbearing potential, a negative urine pregnancy test should be done within 48 hours before the intervention and must use an effective contraceptive method.

Exclusion Criteria:

1. Cardiac surgery contraindications.
2. Patients who require other interventions than the isolated aortic valve replacement or with coronary artery bypass surgery and / or in combination with ascending aorta replacement surgery as concomitant procedure.
3. Patients with LVEF < 30%.
4. Cardiac surgery reintervention.
5. Cardiogenic shock or hemodynamic instability within 24 hours prior to surgery.
6. Patient who are not willing to attend to the required follow-up visit.
7. Patients with active endocarditis (in the case of cured endocarditis, the presence of at least two negative blood cultures must be confirmed before their inclusion in the study).
8. Patient undergoing hemodialysis or with severe renal impairment (eGFR<30ml/min/1,7m2).
9. Pregnant women.
10. Patients with hyperparathyroidism.
11. Life expectancy less than 2 years.
12. Patients with a history or diagnosis of a medical problem or psychiatric illness or disorder that, according to the investigator evaluation, would make the patient not eligible to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Transvalvular gradient | Up to 12 months
  Dokimos Plus aortic valve transvalvular gradient at 6 months and at 12 months after the implantation.

SECONDARY OUTCOMES:
Number of participants with abasence of valve deterioration | 12 months
  Assess the absence of structural valve deterioration (morphological and hemodynamic) after 12 months follow-up.
Number of participants with absence of non-structural valve deterioration | 12 months
  Assess the absence of non-structural valve deterioration after 12 months follow-up.
Number of participants with absence of endocarditis or thrombosis | 10 years
  Asses the absence of endocarditis or thrombosis.
Number of participants with need for prosthetic replacement | 10 years
  Assess the need for prosthetic replacement.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Muñoz, Principal Investigator — Head of Cardiac Surgery Service in the Hospital GT i Pujol, Badalona, Barcelona; Manuel Castellà, Principal Investigator — Head of Cardiac Surgery Service in the Hospital Clínic de Barcelona; Albert Miralles, Principal Investigator — Head of Cardiac Surgery Service in HU. de Bellvitge, Hospitalet de Ll, Barcelona
Locations (3):
- Spain (3):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clínic Barcelona, Barcelona